CLINICAL TRIAL: NCT05494723
Title: A Phase 1 Study of the Safety and Efficacy of YB-1113 in Treatment of Premature Ovarian Insufficiency (POI) Via Intravenous Infusion
Brief Title: Safety and Efficacy of YB-1113 in Treatment of POI
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bright Cell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YB1113-POI
Record Dates: First submitted 2022-08-06; First posted 2022-08-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: POI

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low-dose (Experimental): Low-dose YB-1113
  Interventions: Drug: YB-1113
- High-dose (Experimental): High-dose YB-1113
  Interventions: Drug: YB-1113

INTERVENTIONS:
Drug: YB-1113 — Human umbilical cord tissue-derived mesenchymal stem cells (hUC-MSC)

SUMMARY:
This phase 1 study is to evaluate the safety and tolerability of YB-1113 administered via intravenous (IV) infusion in the treatment of premature ovarian insufficiency (POI).

ELIGIBILITY:
Key Inclusion Criteria:

1. Female, 18 to <40 years old, who are seeking fertility or preservation of fertility
2. Oligo/Amenorrhea for at least 4 months
3. At least two menopausal FSH levels (≥ 25 IU/L) with 4 to 6 weeks interval.
4. AMH levels ≤ 1.0 ng/mL (measured on day 2-5 of the menstrual period).
5. Subjects who are generally healthy by laboratory tests (normal complete blood count (CBC), comprehensive metabolic panel (CMP), and urinalysis) at screening
6. For subjects who had contraception before, the duration of amenorrhea should be more than 3 months after discontinuation of the oral contraception pill (OCP) or more than 6 months after discontinuation of Depo Provera (or similar) therapies

Key Exclusion Criteria:

1. 1. Primary amenorrhea or FSH ≥ 40 IU/L
2. Presence of contraindications to pregnancy
3. POI due to cytotoxic chemotherapy or radiation therapy
4. Subjects with FMR1 premutation (fragile X syndrome), a BMP15 mutation or family history of POI
5. Subjects under hormonal treatments including hormone replacement therapy (HRT) for osteoporosis, cardiovascular disease, or recalcitrant vasomotor symptomatology.
6. Washout period less than 3 months for HRT.
7. Subjects with a history of breast cancer or other estrogen responsive cancer.
8. Subjects with existing malignant neoplasm, under active management for malignant neoplasm or under active surveillance for malignant neoplasm.
9. Subjects with history of thromboembolic events such as pulmonary embolism, stroke, or ischemic heart disease
10. Subjects with uncontrolled hypertension, kidney disease, liver disease, or polycystic ovary syndrome (PCOS)
11. Subjects with endocrinopathies including Cushing's disease, thyroid disease, congenital adrenal hyperplasia and hyperprolactinemia.
12. Subjects under active management for autoimmune disease.
13. Subjects with intra-uterine devices (IUDs).
14. Subjects who are pregnant, breastfeeding, or whose urinary pregnancy test is positive before participation in the study.
15. Subjects who are allergic to low-molecular-weight heparin sodium or human albumin.
16. Subjects with polyglandular autoimmune disease or other conditions require chronic administration of steroids higher than 30 mg/day of hydrocortisone or its equivalent
17. Subjects with hereditary or acquirement coagulopathies, including but not limited to hemophilia, Von Willebrand disease, liver disease, Vitamin K deficiency, and platelet disorders.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-12-09 (Estimated); Primary Completion 2028-01-09 (Estimated); Study Completion 2028-04-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (AE) | 52 weeks
  Reported treatment-related AE and serious adverse events (SAE)

SECONDARY OUTCOMES:
Blood anti-Müllerian hormone (AMH) level | 2, 6, 12, 24, and 52 weeks
  Changes of AMH level from baseline
Follicle-stimulating hormone (FSH) and estradiol (E2) levels | 2, 6, 12, 24, and 52 weeks
  Changes of FSH and E2 from baseline
Antral follicle counts (AFC) | 2, 6, 12, 24, and 52 weeks
  Changes of AFC numbers from baseline

IPD SHARING:
Plan to Share IPD: No